CLINICAL TRIAL: NCT00262938
Title: Lifestyle Change and Quality of Life in Obese Endometrial Cancer Survivors
Brief Title: Lifestyle Change and Quality of Life in Obese Patients With Stage I/II Endometrial Cancer in Remission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5804; NCT00420979 (obsolete NCT alias)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Endometrial Cancer; Weight Changes
Keywords: stage I endometrial carcinoma; stage II endometrial carcinoma; weight changes
MeSH Terms: conditions — Endometrial Neoplasms; Body Weight Changes | interventions — Counseling; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Active Comparator): Patients undergo weekly contact with a dietitian; exercise intervention for 6 months; and physician counseling.Patients undergo quality of life, exercise, and clinical assessments at baseline and at 3, 6, and 12 months.
  Interventions: Behavioral: behavioral dietary intervention; Other: counseling intervention; Other: educational intervention; Other: preventative dietary intervention; Procedure: quality-of-life assessment
- Without Counseling (Active Comparator): Patients undergo quality of life, exercise, and clinical assessments at baseline and at 3, 6, and 12 months.
  Interventions: Procedure: quality-of-life assessment

INTERVENTIONS:
Behavioral: behavioral dietary intervention — Patients undergo weekly contact with a dietitian; exercise intervention for 6 months; and physician counseling at baseline and at 3, 6, and 12 months. Patients undergo quality of life assessments and clinical assessments at baseline and at 3, 6, and 12 months.
  Arms: Lifestyle counseling
Other: counseling intervention — Patients undergo weekly contact with a dietitian; exercise intervention for 6 months; and physician counseling at baseline and at 3, 6, and 12 months. Patients undergo quality of life assessments and clinical assessments at baseline and at 3, 6, and 12 months.
  Arms: Lifestyle counseling
Other: educational intervention — Patients undergo weekly contact with a dietitian; exercise intervention for 6 months; and physician counseling at baseline and at 3, 6, and 12 months. Patients undergo quality of life assessments and clinical assessments at baseline and at 3, 6, and 12 months.
  Arms: Lifestyle counseling
Other: preventative dietary intervention — Patients undergo weekly contact with a dietitian; exercise intervention for 6 months; and physician counseling at baseline and at 3, 6, and 12 months. Patients undergo quality of life assessments and clinical assessments at baseline and at 3, 6, and 12 months.
  Arms: Lifestyle counseling
Procedure: quality-of-life assessment — Patients undergo quality of life assessments and clinical assessments at baseline and at 3, 6, and 12 months.

SUMMARY:
RATIONALE: Exercise and dietary counseling may affect weight loss and improve the quality of life of obese endometrial cancer patients and may help them live longer and more comfortably.

PURPOSE: This randomized clinical trial is studying the effects of exercise and dietary counseling on weight loss and quality of life of obese patients with stage I or stage II endometrial cancer in remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the combined effect of exercise and dietary counseling on the weight loss and quality of life of obese patients with stage I or II endometrial cancer in remission.

Secondary

* Determine the feasibility and acceptability of lifestyle interventions in these patients.

OUTLINE: This is a randomized, controlled study. Patients are stratified according to age and body mass index (25-29.9 vs ≥ 30). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo weekly contact with a dietitian; exercise intervention for 6 months; and physician counseling at baseline and at 3, 6, and 12 months. Patients undergo quality of life assessments and clinical assessments at baseline and at 3, 6, and 12 months.
* Arm II: Patients undergo quality of life, exercise, and clinical assessments at baseline and at 3, 6, and 12 months.

After completion of study treatment, patients are followed at 1 year.

PROJECTED ACCRUAL: Approximately 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed endometrial cancer meeting the following criteria:

  * Stage I or II disease
  * Post-operative total abdominal hysterectomy and bilateral salpingo-oophorectomy
  * Disease in remission
* Body Mass Index (BMI) ≥ 25

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY: Not specified

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-02; Primary Completion 2006-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Quality of life as measured by Functional Assessment of Cancer Therapy for General Cancer (FACT-G) and Functional Assessment of Cancer Therapy for Fatigue (FACT-F) at baseline, 3, 6, and 12 months | baseline, 3, 6, and 12 months
Weight loss as measured by weight, body mass index (BMI), waist circumference, Weight Efficacy Life Style Questionnaire, Three Factor Eating Inventory Questionnaire, and Leisure Score index at baseline, 3, 6, and 12 months | baseline, 3, 6, and 12 months
Functional status as measured by ECOG performance status, and short-form health survey with 36 questions (SF-36) | baseline, 3, 6, and 12 months
Comorbidities as measured by Charlson Co-Morbidity Score at baseline, 3, 6, and 12 months | baseline, 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vivian von Gruenigen, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] von Gruenigen VE, Waggoner SE, Frasure HE, Kavanagh MB, Janata JW, Rose PG, Courneya KS, Lerner E. Lifestyle challenges in endometrial cancer survivorship. Obstet Gynecol. 2011 Jan;117(1):93-100. doi: 10.1097/AOG.0b013e31820205b3. PMID 21173649
- [Derived] von Gruenigen VE, Gibbons HE, Kavanagh MB, Janata JW, Lerner E, Courneya KS. A randomized trial of a lifestyle intervention in obese endometrial cancer survivors: quality of life outcomes and mediators of behavior change. Health Qual Life Outcomes. 2009 Feb 25;7:17. doi: 10.1186/1477-7525-7-17. PMID 19243603